CLINICAL TRIAL: NCT04479358
Title: COVIDOSE-2: A Multi-center, Randomized, Controlled Phase 2 Trial Comparing Early Administration of Low-dose Tocilizumab to Standard of Care in Hospitalized Patients With COVID-19 Pneumonitis Not Requiring Invasive Ventilation
Brief Title: Low-dose Tocilizumab Versus Standard of Care in Hospitalized Patients With COVID-19
Acronym: COVIDOSE-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment of patients into the trial
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-1179
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19; Tocilizumab
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two sub-studies in parallel, each of three arms (maximum).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sub-study A, Tocilizumab-Free Standard of Care (Active Comparator): Patient assigned to Sub-study A by primary treating physicians. Patient enrolled on trial sub-study A and randomized to receive no tocilizumab.
  Interventions: Other: Standard of Care
- Sub-study A, Tocilizumab 40mg (Experimental): Patient assigned to Sub-study A by primary treating physicians. Patient enrolled on trial sub-study A and randomized to receive tocilizumab 40mg.
  Interventions: Drug: Tocilizumab
- Sub-study A, Tocilizumab 120mg (Experimental): Patient assigned to Sub-study A by primary treating physicians. Patient enrolled on trial sub-study A and randomized to receive tocilizumab 120mg.
  Interventions: Drug: Tocilizumab
- Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care (Active Comparator): Patient assigned to Sub-study B by primary treating physicians. Patient enrolled on trial sub-study B and randomized to receive standard of care tocilizumab dose (400mg or 8mgkg).
  Interventions: Other: Standard of Care
- Sub-study B, Tocilizumab 40mg (Experimental): Patient assigned to Sub-study B by primary treating physicians. Patient enrolled on trial sub-study B and randomized to receive standard of care tocilizumab 40mg.
  Interventions: Drug: Tocilizumab
- Sub-study B, Tocilizumab 120mg (Experimental): Patient assigned to Sub-study B by primary treating physicians. Patient enrolled on trial sub-study B and randomized to receive standard of care tocilizumab 120mg.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 40mg
  Other Names: Tocilizumab 40mg
  Arms: Sub-study A, Tocilizumab 40mg; Sub-study B, Tocilizumab 40mg
Drug: Tocilizumab — Tocilizumab 120mg
  Other Names: Tocilizumab 120mg
  Arms: Sub-study A, Tocilizumab 120mg; Sub-study B, Tocilizumab 120mg
Other: Standard of Care — Tocilizumab-Free Standard of Care
  Arms: Sub-study A, Tocilizumab-Free Standard of Care
Other: Standard of Care — Tocilizumab 400mg or 8mg/kg
  Arms: Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care

SUMMARY:
Tocilizumab is an effective treatment for severe coronavirus disease 2019 (Covid-19) pneumonia and related inflammation. Given limited global supplies, clarification of the optimal tocilizumab dose is critical. We conducted an open-label, randomized, controlled trial evaluating two different dose levels of tocilizumab in Covid-19 (40mg and 120mg). Randomization was stratified on remdesivir and corticosteroid at enrollment. The primary outcome was the time to recovery. The key secondary outcome was 28-day mortality.

DETAILED DESCRIPTION:
COVID-19's high mortality may be driven by hyperinflammation. Interleukin-6 (IL-6) axis therapies may reduce COVID-19 mortality. Retrospective analyses of tocilizumab in severe to critical COVID-19 patients have demonstrated survival advantage and lower likelihood of requiring invasive ventilation following tocilizumab administration. The majority of patients have rapid resolution (i.e., within 24-72 hours following administration) of both clinical and biochemical signs (fever and CRP, respectively) of hyperinflammation with only a single tocilizumab dose.

The investigators hypothesized that a dose of tocilizumab significantly lower than the EMA- and FDA-labeled dose (8mg/kg) as well as the emerging standard of care dose (400mg) may be effective in patients with COVID-19 pneumonitis and hyperinflammation. Advantages to the lower dose of tocilizumab may include lower likelihood of secondary bacterial infections as well as extension of this drug's limited supply. The investigators conducted an adaptive single-arm phase 2 trial (NCT04331795) evaluating clinical and biochemical response to low-dose tocilizumab in patients with COVID-19 pneumonitis and hyperinflammation.

This multi-center, prospective, randomized controlled phase 2 trial -- designed as two sub-studies to allow for the possible emergence of data demonstrating the clinical efficacy of tocilizumab 8mg/kg or 400mg -- formally tests the clinical efficacy of low-dose tocilizumab in COVID-19 pneumonia.

Sub-Study A Primary Objective A: To establish whether low-dose tocilizumab reduces the time to clinical recovery in patients with COVID-19 pneumonitis and hyperinflammation, when compared to a tocilizumab-free standard of care.

Hypothesis A: The investigators hypothesize that low-dose tocilizumab, when compared to a tocilizumab-free standard of care, decreases the time to recovery in hospitalized, non-invasively ventilated patients with COVID-19 pneumonitis and hyperinflammation by three days or more.

Sub-Study B Primary Objective B: To establish whether low-dose tocilizumab is near-equivalent to high-dose tocilizumab (400mg or 8 mg/kg) in reducing the time to clinical recovery in patients with COVID-19 pneumonitis and hyperinflammation.

Hypothesis B: The investigators hypothesize that low-dose tocilizumab is near-equivalent to high-dose tocilizumab in reducing the time to clinical recovery in hospitalized, non-invasively ventilated patients with COVID-19 pneumonitis and hyperinflammation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Approval from the patient's primary inpatient service
* Hospitalized
* Fever, documented in electronic medical record and defined as: T ≥ 38 degrees C by any conventional clinical method (forehead, tympanic, oral, axillary, rectal)
* Positive test for active SARS-CoV-2 infection
* Radiographic evidence of infiltrates on chest radiograph (CXR) or computed tomography (CT)
* Ability to provide written informed consent on the part of the subject or, in the absence of decisional capacity of the subject, an appropriate surrogate (e.g. a legally authorized representative).

Exclusion Criteria:

* Concurrent use of invasive mechanical ventilation
* Concurrent use of vasopressor or inotropic medications
* Previous receipt of tocilizumab or another anti-IL6R or IL-6 inhibitor in the year prior.
* Known history of hypersensitivity to tocilizumab.
* Diagnosis of end-stage liver disease or listed for liver transplant.
* Elevation of AST or ALT in excess of 10 times the upper limit of normal.
* Neutropenia (Absolute neutrophil count < 500/uL).
* Thrombocytopenia (Platelets < 50,000/uL).
* On active therapy with a Bruton's tyrosine kinase-targeted agent, which include the following:
* Acalabrutinib
* Ibrutinib
* Zanubrutinib
* On active therapy with a JAK2-targeted agent, which include the following:
* Tofacitinib
* Baricitinib
* Upadacitinib
* Ruxolitinib
* Any of the following biologic immunosuppressive agent (and any biosimilar versions thereof) administered in the past 6 months or less::
* Abatacept
* Adalimumab
* Alemtuzumab
* Atezolizumab
* Belimumab
* Blinatumomab
* Brentuximab
* Certolizumab
* Daratumumab
* Durvalumab
* Eculizumab
* Elotuzumab
* Etanercept
* Gemtuzumab
* Golimumab
* Ibritumomab
* Infliximab
* Inotuzumab
* Ipilimumab
* Ixekizumab
* Moxetumomab
* Nivolumab
* Obinutuzumab
* Ocrelizumab
* Ofatumumab
* Pembrolizumab
* Polatuzumab
* Rituximab
* Rituximab
* Sarilumab
* Secukinumab
* Tocilizumab
* Tositumumab
* Tremelimumab
* Urelumab
* Ustekinumab
* History of bone marrow transplantation (including chimeric antigen receptor T-cell) or solid organ transplant
* Known history of Hepatitis B or Hepatitis C (patients who have completed curative-intent anti-HCV treatments are not excluded from trial)
* Positive result on hepatitis B or C screening
* Known history of mycobacterium tuberculosis infection at risk for reactivation
* Known history of gastrointestinal perforation
* Active diverticulitis
* Multi-organ failure as determined by primary treating physicians
* Any other documented serious, active infection besides COVID-19 - including but not limited to: lobar pneumonia consistent with bacterial infection, bacteremia, culture-negative endocarditis, or current mycobacterial infection - at the discretion of primary treating physicians
* Pregnant patients or nursing mothers
* Patients who are unable to discontinue scheduled antipyretic medications, either as monotherapy (e.g., acetaminophen or ibuprofen [aspirin is acceptable]) or as part of combination therapy (e.g., hydrocodone/acetaminophen, aspirin/acetaminophen/caffeine [Excedrin®])
* CRP < 40 mg/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankti D Reid, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of this article, after de-identification. Sharing period will be 1 month after data are published and available indefinitely thereafter. Researchers who provide methodologically sound proposals for the purposes of achieving stated aims in their proposal will be eligible for data-sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: From 1 month following publication of data. Available indefinitely thereafter.
Access Criteria: Proposals will need to be sent to study principal investigators. Requestors will need to sign a data access request form. Link to be determined.

REFERENCES:
- [Background] Strohbehn GW, Reid PD, Ratain MJ. Applied Clinical Pharmacology in a Crisis: Interleukin-6 Axis Blockade and COVID-19. Clin Pharmacol Ther. 2020 Sep;108(3):425-427. doi: 10.1002/cpt.1931. Epub 2020 Jul 4. PMID 32488861

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sub-study A, Tocilizumab-Free Standard of Care | Sub-study A, Tocilizumab 40mg | Sub-study A, Tocilizumab 120mg | Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care | Sub-study B, Tocilizumab 40mg | Sub-study B, Tocilizumab 120mg
Started | 26 | 25 | 26 | 3 | 3 | 2
Completed | 26 | 25 | 25 | 3 | 3 | 1
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-study A, Tocilizumab-Free Standard of Care | Sub-study A, Tocilizumab 40mg | Sub-study A, Tocilizumab 120mg | Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care | Sub-study B, Tocilizumab 40mg | Sub-study B, Tocilizumab 120mg | Total
Number analyzed (Participants) | 26 | 25 | 25 | 3 | 3 | 1 | 83
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [27 to 97] | 56.5 [31 to 82] | 59.2 [30 to 95] | 49.7 [39 to 60] | 53.3 [24 to 80] | 72 [72 to 72] | 57.5 [24 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 15 | 3 | 2 | 1 | 45
  Male | 17 | 10 | 10 | 0 | 1 | 0 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 23 | 21 | 23 | 3 | 2 | 1 | 73
  White | 1 | 3 | 2 | 0 | 1 | 0 | 7
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 25 | 3 | 3 | 1 | 83

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery
Description: Day of recovery is defined as the first day on which the patient achieves one of the following two categories from the seven-point ordinal scale: 6) Hospitalized, not requiring supplemental oxygen or ongoing medical care or 7) Not hospitalized. Time to recovery is the number of days from randomization to achievement of this status. Note that the ordinal scale is measured once daily, with the patient's worst clinical status during the 24-hour time period (0:00-23:59) being documented.
Time Frame: 28 days
Population: Note: for confidence intervals below, -9999 and 9999 = Upper or lower limit cannot be estimated due to insufficient number of participants with events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sub-study A, Tocilizumab-Free Standard of Care | Sub-study A, Tocilizumab 40mg | Sub-study A, Tocilizumab 120mg | Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care | Sub-study B, Tocilizumab 40mg | Sub-study B, Tocilizumab 120mg
Number analyzed (Participants) | 26 | 25 | 25 | 3 | 3 | 1
days | 5 [4 to 6] | 7 [4 to 9] | 4 [4 to 5] | 7 [2.4 to NA] — Insufficient number of patients to compute upper confidence limit | 6 [4 to NA] — Insufficient number of patients to compute upper confidence limit | 8 [NA to NA] — Insufficient number of patients to compute confidence limits

2. Secondary Outcome: Achievement of Recovery
Description: This will be defined as the percentage of patients in a given arm of the study achieving one of the above two categories on the ordinal scale on day 7. Note that the ordinal scale is measured once daily, with the patient's worst clinical status during the 24-hour time period (0:00-23:59) being documented.
Time Frame: 7 days
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: This will be defined as the percentage of patients in a given arm of the study who are alive thirty days following randomization. Patients who are discharged to hospice will be counted as deceased on the day of discharge. Patients who are transitioned to inpatient hospice or inpatient comfort measures only will be counted as deceased on the day of transition.
Time Frame: 28 days
Reporting Status: Not Posted

4. Secondary Outcome: Hospital Length of Stay
Description: This will be defined as the number of days that pass between the day of a patient's randomization and his or her discharge from the hospital.
Time Frame: Up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Response: Maximum Temperature (Tmax) Response
Description: Maximum temperature within 24-hour periods of time immediately prior to, immediately following, and then every 24 hours thereafter randomization. The primary endpoint is a measured Tmax in the 24-hour period immediately following randomization that is lower than the measured Tmax in the 24-hour period immediately preceding randomization.
Time Frame: 24 hours
Reporting Status: Not Posted

6. Secondary Outcome: Clinical Response: Rate of Non-Elective Invasive Mechanical Ventilation
Description: This will be a binary outcome defined as worsening COVID-19 disease resulting in the use of invasive mechanical ventilation during the course of the patient's COVID-19 infection.
Time Frame: Up to 28 days
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Response: Duration of Non-Elective Invasive Mechanical Ventilation
Description: This will be a continuous outcome defined by the amount of time between initiation and cessation of non-elective invasive mechanical ventilation.
Time Frame: Up to 28 days
Reporting Status: Not Posted

8. Secondary Outcome: Clinical Response: Time to Non-Elective Invasive Mechanical Ventilation
Description: This will be a continuous outcome defined by the amount of time between randomization and the initiation of non-elective invasive mechanical ventilation. This will be treated as a time-to-event with possible censoring.
Time Frame: Up to 28 days
Reporting Status: Not Posted

9. Secondary Outcome: Clinical Response: Rate of Vasopressor/Inotrope Utilization
Description: This will be a binary outcome defined as utilization of any vasopressor or inotropic medication.
Time Frame: Up to 28 days
Reporting Status: Not Posted

10. Secondary Outcome: Clinical Response: Duration of Vasopressor/Inotrope Utilization
Description: This will be a continuous outcome defined by the amount of time between initiation of first and cessation of last vasopressor medications.
Time Frame: Up to 28 days
Reporting Status: Not Posted

11. Secondary Outcome: Clinical Response: Time to Vasopressor/Inotrope Utilization
Description: This will be a continuous outcome defined by the amount of time between randomization and the initiation of any vasopressor or inotropic medication. This will be treated as a time-to-event with possible censoring.
Time Frame: Up to 28 days
Reporting Status: Not Posted

12. Secondary Outcome: Clinical Response: Duration of Increased Supplemental Oxygen From Baseline
Description: This will be an ordinal outcome defined by the number of days counted from randomization over which the participant requires supplemental oxygen in excess over his/her baseline supplemental oxygen requirement. The supplemental oxygen requirement is defined as the highest liters-per-minute flow of supplemental oxygen required by the patient each day over the course of the hospitalization.
Time Frame: 28 days
Reporting Status: Not Posted

13. Secondary Outcome: Biochemical Response: C-reactive Protein Response Rate
Description: This will be a binary outcome defined as the presence or absence of a decline in CRP of ≥ 25% from baseline CRP in the 27 +/- 3 hours after tocilizumab administration, as compared to pre-treatment baseline.
Time Frame: 24 hours
Reporting Status: Not Posted

14. Secondary Outcome: Safety: Rate of Secondary Infection
Description: This will be defined as the percentage of patients in a study arm who develop serious non-COVID-19 viral, bacterial, or fungal infections (e.g., bloodstream infection, hospital-acquired pneumonia, ventilator-associated pneumonia, opportunistic infection) following randomization and up to the 28-day assessment of overall survival.
Time Frame: 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Sub-study A, Tocilizumab-Free Standard of Care | Sub-study A, Tocilizumab 40mg | Sub-study A, Tocilizumab 120mg | Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care | Sub-study B, Tocilizumab 40mg | Sub-study B, Tocilizumab 120mg
All-Cause Mortality (participants affected / at risk) | 1/26 | 3/25 | 0/25 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25 | 0/25 | 0/3 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 23/26 | 22/25 | 21/25 | 3/3 | 3/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sub-study A, Tocilizumab-Free Standard of Care (N=26) | Sub-study A, Tocilizumab 40mg (N=25) | Sub-study A, Tocilizumab 120mg (N=25) | Sub-study B, Tocilizumab 400mg or 8mg/kg Standard of Care (N=3) | Sub-study B, Tocilizumab 40mg (N=3) | Sub-study B, Tocilizumab 120mg (N=1)
Anemia (Blood and lymphatic system disorders) | 3 | 6 | 3 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 6 | 8 | 5 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0 | 0 | 0
Cardiac disorders - other (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 0
General disorders and administration site conditions (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 0 | 0
Infections and infestations (Infections and infestations) | 1 | 2 | 2 | 0 | 0 | 0
Alanine aminotransferase (Investigations) | 9 | 12 | 7 | 1 | 0 | 1
Aspartate aminotransferase (Investigations) | 9 | 12 | 5 | 2 | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 3 | 4 | 0 | 0 | 1
Investigations - other (Investigations) | 15 | 13 | 13 | 1 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 0 | 0
Renal and urinary disorders - other (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 6 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 1 | 2 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT04479358/Prot_SAP_000.pdf